CLINICAL TRIAL: NCT05947175
Title: The Vertebral Bone Marrow Clot as Autologous Cell-therapy and Multifunctional Bio-scaffold Targeting the Key Challenges for Spinal Fusion Surgery
Brief Title: Vertebral Bone Marrow Clot for Spinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MORE_FOR_SPINE
Record Dates: First submitted 2023-06-27; First posted 2023-07-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Degenerative Spine Diseases
Keywords: Spine; Spinal fusion; Degenerative diseases; Vertebral bone marrow; Clot
MeSH Terms: interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group - vertebral bone marrow (vBMA) clot (Experimental): Bone allograft chips will be obtained from Istituto Ortopedico Rizzoli while vBMA will be harvested from each patient vertebral pedicle with the preparation of the site for pedicle screw insertion during spinal surgery. After the positioning of pedicle screws, the decompression of the cauda and nerve roots will be achieved with a hemilaminectomy and foraminotomy. vBMA clot associated with bone allograft chips will be opposed on the hemi-laminae and transvers process on the contralateral side of the hemilaminectomy. On the hemilaminectomy side, foramino-arthrectomy will be performed to insert the interbody fusion cage if necessary. After aspiration, the vBMA will be clotted and used for surgical procedure. vBMA clot associated to bone allograft chips will be applied on each side of the vertebra according to the number of segments to be fused.
  Interventions: Biological: Vertebral bone marrow (vBMA) clot
- Control - bone allograft chips (Active Comparator): Bone allograft chips will be obtained from Istituto Ortopedico Rizzoli. In detail, conventional posterior approach for lumbar SF will be performed. After the positioning of pedicle screws, the decompression of the cauda and nerve roots will be achieved with a hemilaminectomy and foraminotomy. Bone allograft chips alone will be opposed on the hemi-laminae and transvers process on the contralateral side of the hemilaminectomy. On the hemilaminectomy side, foramino-arthrectomy will be performed to insert the interbody fusion cage if necessary.
  Interventions: Other: Bone allograft chips

INTERVENTIONS:
Biological: Vertebral bone marrow (vBMA) clot — The clotted vBMA will be obtained from vertebral bone marrow aspirate.The vBMA clot contain mesenchymal stem cells (MSCs), growth factors, platelet and osteogenic and anti-inflammatory mediators.
  Arms: Experimental group - vertebral bone marrow (vBMA) clot
Other: Bone allograft chips — Bone allograft chips will be obtained from Musculoskeletal Tissue Bank at IRCCS Istituto Ortopedico Rizzoli.
  Arms: Control - bone allograft chips

SUMMARY:
Spinal fusion (SF) is a common orthopedic procedure to treat spinal diseases. Apart from fixation systems, the procedure requires bone grafting to further improve SF. Cell-based therapies as vertebral bone marrow aspirate (vBMA) with bone allograft were developed as alternative to bone autograft in SF. However, vBMA use is limited by the lack of a standardized procedure, of a structural texture and by the possibility of diffusion away from the implant site. Recently, the potential use of a new formulation of vBMA, named vBMA clot, has been described. The project aims at evaluating the clinical evidence and the biological features of vBMA clot associated to bone allograft for SF surgery, considering age and gender related differences. A randomized controlled trial will prove the efficacy of the treatment and advanced preclinical studies will improve the knowledge on vBMA clot regenerative and anti-inflammatory properties, exploring for the first time its antibacterial characteristics.

DETAILED DESCRIPTION:
To evaluate the efficacy of autologous vBMA clot in SF procedures in patients with degenerative spine diseases, a randomized controlled trial (RCT) will be carried out. The study will compare patients treated with autologous vBMA clot associated to bone allograft chips versus bone allograft chips alone (standard treatment), also evaluating whether patient age and gender are associated with differences in the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* degenerative spinal disorders (based radiological diagnosis)
* posterior spinal stabilization ≤ 5 levels
* age between 18-80 years at the time of surgery

Exclusion Criteria:

* HIV
* HBV
* HCV
* coagulations disorders
* pregnant or breast-feeding women
* cancer
* infections
* previous spinal surgery
* radio- chemotherapy
* myeloproliferative disease
* chronic steroid medication, thyroxin, immunodepression

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Brantigan classification | At baseline (day 0)
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at 1, 3, 6, 12 months of FU, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).
Brantigan classification | 1 month
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at 1, 3, 6, 12 months of FU, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).
Brantigan classification | 3 months
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at 1, 3, 6, 12 months of FU, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).
Brantigan classification | 6 months
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at 1, 3, 6, 12 months of FU, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).
Brantigan classification | 12 months
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at 1, 3, 6, 12 months of FU, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).

SECONDARY OUTCOMES:
Re-operation rate | At baseline (day 0)
  The radiological outcome is the reduction of re-operation rate due to pseudoarthrosis that will be estimate by Brantigan classification.
Re-operation rate | 1 month
  The radiological outcome is the reduction of re-operation rate due to pseudoarthrosis that will be estimate by Brantigan classification.
Re-operation rate | 3 month
  The radiological outcome is the reduction of re-operation rate due to pseudoarthrosis that will be estimate by Brantigan classification.
Re-operation rate | 6 month
  The radiological outcome is the reduction of re-operation rate due to pseudoarthrosis that will be estimate by Brantigan classification.
Re-operation rate | 12 month
  The radiological outcome is the reduction of re-operation rate due to pseudoarthrosis that will be estimate by Brantigan classification.
Visual Analogue Score | At baseline (day 0)
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Visual Analogue Score | 1 month
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Visual Analogue Score | 3 months
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Visual Analogue Score | 6 months
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Visual Analogue Score | 12 months
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Oswestry Disability Index | At baseline (day 0)
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
Oswestry Disability Index | 1 month
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
Oswestry Disability Index | 3 months
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
Oswestry Disability Index | 6 months
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
Oswestry Disability Index | 12 months
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
Short Form Health Survey 36 | At baseline (day 0)
  Short Form Health Survey 36 (SF-36) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)
Short Form Health Survey 36 | 1 month
  Short Form Health Survey 36 (SF-36) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)
Short Form Health Survey 36 | 3 months
  Short Form Health Survey 36 (SF-36) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)
Short Form Health Survey 36 | 6 months
  Short Form Health Survey 36 (SF-36) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)
Short Form Health Survey 36 | 12 months
  Short Form Health Survey 36 (SF-36) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salamanna F, Contartese D, Giavaresi G, Sicuro L, Barbanti Brodano G, Gasbarrini A, Fini M. A Rationale for the Use of Clotted Vertebral Bone Marrow to Aid Tissue Regeneration Following Spinal Surgery. Sci Rep. 2020 Mar 5;10(1):4115. doi: 10.1038/s41598-020-60934-2. PMID 32139727
- [Result] Salamanna F, Contartese D, Nicoli Aldini N, Barbanti Brodano G, Griffoni C, Gasbarrini A, Fini M. Bone marrow aspirate clot: A technical complication or a smart approach for musculoskeletal tissue regeneration? J Cell Physiol. 2018 Apr;233(4):2723-2732. doi: 10.1002/jcp.26065. Epub 2017 Jul 24. PMID 28639702
- [Result] Salamanna F, Contartese D, Borsari V, Pagani S, Barbanti Brodano G, Griffoni C, Ricci A, Gasbarrini A, Fini M. Two Hits for Bone Regeneration in Aged Patients: Vertebral Bone Marrow Clot as a Biological Scaffold and Powerful Source of Mesenchymal Stem Cells. Front Bioeng Biotechnol. 2022 Jan 18;9:807679. doi: 10.3389/fbioe.2021.807679. eCollection 2021. PMID 35118056
- [Derived] Sartori M, Tedesco G, Spinnato P, Mazzotti A, Gasbarrini A, Faldini C, Miceli M, Giavaresi G, Salamanna F. The Vertebral Bone Marrow clot as cell therapy and multifunctional bioscaffold for spinal fusion surgery: protocol for a randomized clinical trial. Front Med (Lausanne). 2025 May 9;12:1591041. doi: 10.3389/fmed.2025.1591041. eCollection 2025. PMID 40417680